CLINICAL TRIAL: NCT00150098
Title: Project UNITY - A Randomized Trial of Enhanced HIV Risk Reduction and Vaccine Education Interventions in Reducing Sexual Risk and Increasing Vaccine Trial Knowledge Among HIV-negative, High-risk Women Who Use Non-injection Drugs
Brief Title: Project UNITY - HIV Risk Reduction and Vaccine Education Interventions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York Blood Center (Other)
Collaborators: The New York Academy of Medicine (Other); Rutgers University (Other)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: IRB 406-04; 5R01DA017482-03 (NIH)
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Last update posted 2014-04-08 (Estimated); Status verified 2014-04

CONDITIONS: HIV Infections; Hepatitis B
Keywords: HIV; vaccines; women; substance use
MeSH Terms: conditions — HIV Infections; Hepatitis B; Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- lifestyle counselling (Experimental): Education
  Interventions: Behavioral: Enhanced HIV risk reduction and HIV vaccine education

INTERVENTIONS:
Behavioral: Enhanced HIV risk reduction and HIV vaccine education

SUMMARY:
To determine the efficacy of an enhanced HIV risk reduction intervention delivered concurrently with a vaccination schedule to reduce the number of unprotected vaginal and anal sex acts among HIV-negative, high-risk non-injection drug-using (NIDU) women. To determine the efficacy of an enhanced vaccine education intervention delivered at baseline to increase vaccine knowledge and understanding of a potential HIV vaccine among HIV-negative, high-risk NIDU women.

DETAILED DESCRIPTION:
We are currently screening women (approximately 535) from whom we expect 400 HIV-negative high-risk, non-pregnant NIDU women will be enrolled to participate in a two-arm randomized trial of an enhanced HIV risk reduction intervention plus an enhanced vaccine education intervention compared to controls. At screening, women complete an assessment, receive HIV and HBV pre-test counseling, and are tested for HIV antibody, markers of hepatitis B virus (HBV) infection and pregnancy. At the enrollment visit (2 weeks later), eligible and willing participants are randomized to receive either the enhanced HIV risk reduction intervention plus the enhanced vaccine education intervention or control conditions. Enrolled women provide urine for pregnancy testing. Enrolled women found to be susceptible to HBV are offered hepatitis B (HB) vaccine at the enrollment visit. Follow-up visits coincide with the HB vaccine schedule (1 and 6 months post enrollment) for all women, regardless of whether or not they received HB vaccine. Pregnancy testing is conducted at these follow-up visits. Participants provide sera for HIV antibody testing at the 6- and 12-months visits. A final visit will occur at 12 months post enrollment to assess longer term effects on risk behaviors and knowledge and understanding of vaccine concepts. All standardized interviews are conducted using Audio Computer Assisted Self-Interview (ACASI) technology.

The enhanced HIV risk reduction intervention is a series of three, interactive, individually-delivered, counseling sessions. The enhanced sessions also include tailored male and female condom demonstrations to build skills, and each session concludes with a client-initiated sexual risk reduction goal. The follow-up sessions (at 1 and 6 months) resume by reviewing goal attainment, exploring the reasons and beliefs associated with progress toward that goal. The control group receives the client-centered HIV counseling based on the Centers for Disease Control and Prevention (CDC) Project RESPECT model. Both the control and enhanced risk reduction counseling are delivered at the baseline (time 0) and at follow up visits (1 month and 6 months).

The enhanced vaccine education component will test the two-session model informed consent process outlined by Coletti et al but enhanced with simplified illustrated educational material delivered through flipcharts, video and individual counseling at baseline and 1 week later. The control condition is based on the Coletti two-session informed consent process.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years of age;
* non-injecting use of heroin, cocaine or crack cocaine in the last six months;
* unprotected vaginal sex in the last three months;
* test HIV antibody negative;
* agree to provide specimens for testing (HIV, HBV and pregnancy) and be willing to learn the results of these tests;
* ability to understand spoken English or Spanish;
* agree to be randomized;
* willing to return for visits at 1, 6, and 12 months post-enrollment;
* willing and able to provide informed consent.

Exclusion Criteria:

* history of injection drug use in the previous 3 years;
* pregnant;
* intending to become pregnant in the next 12 months.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2005-02; Primary Completion 2009-11 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
- an HIV risk score, the Vaginal Episode Equivalent (VEE) | approved prior to 12-1-12
- understanding assessment for HIV vaccines. | approved prior to 12-1 2012

SECONDARY OUTCOMES:
-frequency of use of specific drugs | approved prior to 12-1-12
-knowledge of HB vaccine acceptance of hepatitis B vaccine among those susceptible | approved prior to 12-1-12
-adherence to hepatitis B vaccination schedule | approved prior to 12-1-12
-willingness to participate in HIV vaccine trials | approved prior to 12-1-12
-measures of motivators and barriers to receiving hepatitis B vaccine and a candidate HIV vaccine | approved prior to 12-1-12
-incidence of pregnancy | approved prior to 12-1-12

CONTACTS AND LOCATIONS:
Overall Officials: Beryl A Koblin, Ph.D., Principal Investigator — New York Blood Center
Locations (2):
- United States (2):
  - New York Blood Center, New York, New York
  - New York Blood Center - Project Achieve, The Bronx, New York

REFERENCES:
- [Derived] Koblin BA, Bonner S, Hoover DR, Xu G, Lucy D, Fortin P, Putnam S, Latka MH. A randomized trial of enhanced HIV risk-reduction and vaccine trial education interventions among HIV-negative, high-risk women who use noninjection drugs: the UNITY study. J Acquir Immune Defic Syndr. 2010 Mar;53(3):378-87. doi: 10.1097/QAI.0b013e3181b7222e. PMID 20190585